CLINICAL TRIAL: NCT04833231
Title: The Relationship Between Renal Functions and Multi Drug Resistant Organisms in Patients With Ventilator Associated Pneumonia
Brief Title: The Relationship Between Renal Functions and Multi Drug Resistant Organisms
Status: Completed | Type: Observational
Sponsor: Konya Numune Hospital (Other Government)
Responsible Party: Principal Investigator, Omur ILBAN, Principal investigator, Konya Numune Hospital
Other Study IDs: omurilban1
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease; Glomerular Filtration Rate; Drug Resistance
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High eGFR group (eGFR ≥60 mL/ min/1.73 m2): Patients with estimated glomerular filtration rate (eGFR) ≥60 mL/ min/1.73 m2 as high eGFR group
- Low eGFR group (eGFR <60 mL/min/1.73 m2): Patients with estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 as low eGFR group

SUMMARY:
Ventilator-associated pneumonia (VAP) is the most common nosocomial infection in patients receiving invasive mechanical ventilation (MV). Antibiotic resistance poses an increasing threat due to the rise of infections caused by multidrug-resistant organisms (MDROs).Despite the increase in the frequency of MDRO colonisation and infection in dialysis patients, it is not known enough whether the risk of multi-drug resistant (MDR) pneumonia increases in mild-to-severe chronic kidney disease (CKD) (eGFR <60 mL/min/1.73 m2) patients not receiving dialysis. Therefore, in our study, the investigators aimed to evaluate the relationship between renal functions and MDR VAP risk and the specific microbial pattern.

DETAILED DESCRIPTION:
This prospective observational study was performed on adult patients intubated and receiving MV for at least 48 hours in the 42-bed surgical and medical Intensive Care Unit. The study was conducted between August 2019 and January 2021 and approved by the Ethics Committee of Necmettin Erbakan University Medical School. Informed consents were obtained from patients participating in the study or from their relatives. The characteristics of patients with MDRO infection associated with different eGFR categories in VAP patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age and above
* A clinical suspicion of VAP as defined in the American Thoracic Society (ATS) guidelines
* A Clinical Pulmonary Infection Score (CPIS) > 6
* No signs and symptoms of infection at the time of admission to the ICU

Exclusion Criteria:

* Acute kidney injury
* Renal replacement treatment (RRT)
* Dialysis
* Renal transplantation
* Active tuberculosis
* Malnutrition
* Immunosuppression (neutropenia, HIV positivity, transplantation, prednisone treatment of ≥20 mg/day, etc.)
* Any extrapulmonary infection other than VAP at the time of being included in the study
* Respiratory cultures presented fungal agents
* Normal flora
* No growth

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were intubated endotracheally and received mechanical ventilation treatment for at least 48 hours in ICU.
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Multi-drug resistant (MDR) pneumonia | 18 months
  The presence of an infection with a resistant pathogen in patients with impaired renal function (eGFR <60 mL/min/1.73 m2) served as our primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Omur ILBAN, MD, Principal Investigator — Konya Numune Hospital, Department of Intensive Care
Locations (1):
- Konya Numune Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided